CLINICAL TRIAL: NCT06974760
Title: A Prospective, Multicenter, Blinded, Randomized Controlled Clinical Trial to Evaluate the Safety and Efficacy of IVUS Console and IVUS Catheter in Coronary Intervention Procedures
Acronym: IVUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Medical Imaging Technology (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BD-IVUS-002
Record Dates: First submitted 2025-04-16; First posted 2025-05-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Percutaneous Coronary Intervention (PCI); Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Boston IVUS (Other)
  Interventions: Device: IVUS
- Pluse IVUS (Other)
  Interventions: Device: IVUS

INTERVENTIONS:
Device: IVUS — The Participants will receive IVUS examinations from Pulse and Boston

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of IVUS Console and IVUS Catheter in coronary intervention therapy

Participants will:

Undergo IVUS examinations from two different manufacturers（from Pulse and Boston Scientific）

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥ 18 years old;
2. Subjects who require coronary artery intravascular ultrasound (IVUS) guidance prior to stent implantation upon clinical judgment;
3. Subjects who are able to understand and willing to sign the informed consent form (ICF).

Exclusion Criteria:

1. Subjects who are not suitable for percutaneous coronary stent implantation;
2. Subjects who are diagnosed with coronary artery spasm;
3. Subjects with a history of allergy to contrast agents;
4. Subjects who are participating in other clinical trials and have not yet reached the primary endpoint;
5. Subjects who are deemed ineligible to be included in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Effectiveness | From enrollment to the end of treatment at one week
  Measure the Mean Stent Area in square millimeter(MSA)
  Comparison between the MSA measured by the Pulse and Boston Scientific Intravascular Ultrasound Diagnostic System, including mean relative deviation, confidence interval and standard deviation, as assessed by Bland-Altman analysis .

SECONDARY OUTCOMES:
Minimal Lumen Area in square millimeter(MLA) | Estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Comparison between the MLA measured by the Pubmed Intravascular Ultrasound Diagnostic System and Boston Scientific Intravascular Ultrasound Diagnostic System, as assessed by Bland-Altman analysis and Pearson analysis.
Stent Length in millimeter (SL) | Estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Comparison between the SL measured by the Pubmed Intravascular Ultrasound Diagnostic System and Boston Scientific Intravascular Ultrasound Diagnostic System, as assessed by Bland-Altman analysis and Pearson analysis.
The rate of detected stent malapposition, tissue prolapse and dissection | Estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Detection rate of poor adherence, tissue prolapse and intercalation, for each system individually, and comparison between the two systems.
Identification plaque properties | Estimated 1 month on average, by a third-party corelab IVUS image post-analysis
  Rates of lipid-rich plaque, fibrous plaque and calcified plaque, discerned by each system individually, and comparison between the two systems
Stability of system(questionnaire) | estimated 1week on average, by opeartor's rating on questionaire
  Evaluate the stability, ease of use, and clarity of captured images of the both IVUS systems from all enrolled case. Each performance includes three options: excellent, good, and poor.
Maneuvering performance of catheter(questionnaire) | estimated 1week on average, by opeartor's rating on questionaire
  Evaluate the maneuvering performance of catheters in the two systems concluded from all enrolled case, including below measures :the pushability，the crossability and the angiographic visibility，Each performance includes three options: excellent, good, and poor.

OTHER OUTCOMES:
Rate of intraoperative adverse effects | From enrollment to the end of treatment at one weeks
  Rate of device-related adverse effects, for each system individually, and comparison between the two systems.
Rate of successful use of instruments | From enrollment to the end of treatment at one weeks
  Device success rate, defined as a valid IVUS image for each system, and comparison between the two systems

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Anzhen Hospital. Capital Medical University, Beijing
  - The Sixth Medical Center of PLA General Hospital, Beijing
  - Shanghai Tongji Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No